CLINICAL TRIAL: NCT00966186
Title: The 90-degree Rotational Insertion Technique for the Large Size ProSeal Laryngeal Mask Airway
Brief Title: The Rotational Insertion Technique for ProSeal Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jung-won Hwang, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: jungwon
Record Dates: First submitted 2009-08-20; First posted 2009-08-26 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-07

CONDITIONS: General Anesthesia; Elective Surgery
Keywords: ProSeal Laryngeal Mask Airway; Rotational technique; Success rate; Postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard technique (Active Comparator): Proseal laryngeal mask airway was inserted according to the manufacture's instruction manual (insertion with help of index finger insertion)
  Interventions: Procedure: Insertion fo ProSeal laryngeal mask airway
- Rotational technique (Experimental): The entire cuff of the PLMA was placed in the mouth without finger insertion in a midline approach and was rotated 90 degrees counterclockwise around the tongue. The PLMA was then advanced and rotated back until resistance was fel
  Interventions: Procedure: Insertion fo ProSeal laryngeal mask airway

INTERVENTIONS:
Procedure: Insertion fo ProSeal laryngeal mask airway — Insertion fo ProSeal laryngeal mask airway using each of Standard technique or Rotational technique

SUMMARY:
The purpose of this study is to compare two insertion techniques of large size ProSeal laryngeal mask airway. We hypothesized that insertion of ProSeal laryngeal mask airway with 90-degree rotation would reduce the contact surface between the device and pharyngeal wall and make it easy to advance the device over the smooth angle against the posterior pharyngeal wall.We compared the success rate and incidence of complication of the standard technique with the rotational technique.

DETAILED DESCRIPTION:
ProSeal laryngeal mask airway is not easy to be inserted due to its larger cuff especially in Asian population. First-time insertion success rate was lower and more time was required to achieve an effective airway even in well-trained physician. A number of techniques have been described to improve the insertion success rate. However, these techniques are only recommended to be used as backup when the digital or introducer tool techniques fail. We hypothesized that insertion of ProSeal laryngeal mask airway with 90-degree rotation would reduce the contact surface between the device and pharyngeal wall and make it easy to advance the device over the smooth angle against the posterior pharyngeal wall.We compared the success rate and incidence of complication of the standard technique with the rotational technique.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-II

Exclusion Criteria:

* Predicted difficult airway
* Mouth opening less than 2.5 cm
* Present sore throat
* High risk of aspiration

Ages: 27 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-won Hwang, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Jeon YT, Na HS, Park SH, Oh AY, Park HP, Yun MJ, Kim JH, Hwang JW. Insertion of the ProSeal laryngeal mask airway is more successful with the 90 degrees rotation technique. Can J Anaesth. 2010 Mar;57(3):211-5. doi: 10.1007/s12630-009-9241-4. Epub 2010 Jan 15. PMID 20077171

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Technique: Proseal laryngeal mask airway was inserted according to the manufacture's instruction manual
Period: Overall Study
Arm/Group | Standard Technique | Rotational Technique
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Technique | Rotational Technique | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 56 | 108
  >=65 years | 8 | 4 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 49.6 (12.9) | 47.4 (10.7) | 48.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 37 | 38 | 75
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Success of Insertion at First Attempt
Time Frame: 5 minute
Measure: Number; unit: participants
Arm/Group | Standard Technique | Rotational Technique
Number analyzed (Participants) | 60 | 60
participants | 50 | 60

2. Secondary Outcome: Insertion Time, Sealing Pressure and Complication
Time Frame: 5 min - 4 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Standard Technique | Rotational Technique
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
First, as the PLMAs were inserted by two anesthesiologists who were experts in PLMA insertion, these results may not apply to novices. Second, the insertion technique was impossible to blind the anesthesiologists, which might be a source of bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No